CLINICAL TRIAL: NCT02516098
Title: A Single Center, Single-dose, Double-blind, Randomized, Two Period Crossover, Two Stage Design to Determine Bioequivalence of Two Formulations Containing Hyoscine Butylbromide 10mg Sugar Coated Tablets, Under Fasting Conditions
Brief Title: Determine the Bioequivalence of Two Formulations of Hyoscine Butylbromide.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202.850
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — Butylscopolammonium Bromide

ARMS (2):
- Hyoscine butylbromide SCT (Active Comparator)
  Interventions: Drug: hyoscine butylbromide
- Hyoscine butylbromide (Experimental)
  Interventions: Drug: hyoscine butylbromide

INTERVENTIONS:
Drug: hyoscine butylbromide

SUMMARY:
Determine bioequivalence of two forumulations with hyoscine butylbromide 10mg sugar coated tablets.

ELIGIBILITY:
Inclusion criteria:

healthy males and females, aged 18-50years, BMI 18,5-30

Exclusion criteria:

History of hypersensitivity or allergy to IMP

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Bloemfontein, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects who meet the inclusion criteria will be considered eligible to participate in the study. Subjects who meet one or more of the exclusion criteria will not be considered eligible to participate in the study.
Groups:
- REF-T: The subjects received the reference treatment (REF) which was 20 milligram (mg) of hyoscine butylbromide (trade name: Buscopan®, 2*10mg) followed by a washout period of 7 to 14 days followed by the test treatment (T) which was 20 mg of hyoscine butylbromide (trade name: Buscapina®, 2*10mg) followed by a washout period of 7 to 14 days.
  All medications were administered as a single oral dose in the fasted state via a sugar coated tablet.
- T-REF: The subjects received test treatment (T) which was 20 milligram (mg) of hyoscine butylbromide (trade name: Buscapina®, 2*10mg) followed by a washout period of 7 to 14 days followed by the reference treatment (REF) which was 20 mg of hyoscine butylbromide (trade name: Buscopan®, 2*10mg) followed by a washout period of 7 to 14 days.
  All medications were administered as a single oral dose in the fasted state via a sugar coated tablet.
Period: Period 1
Arm/Group | REF-T | T-REF
Started | 28 | 28
Completed | 27 | 28
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Washout After Period 1
Arm/Group | REF-T | T-REF
Started | 27 | 28
Completed | 27 | 27
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | REF-T | T-REF
Started | 27 | 27
Completed | 27 | 26
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout After Period 2
Arm/Group | REF-T | T-REF
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least a single dose of the study medication were included in the safety population (safety population = 56 subjects).
Groups:
- Total: Total of all reporting groups
Arm/Group | REF-T | T-REF | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (7.17) | 24.5 (3.90) | 25.6 (5.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration of Hyoscine Butylbromide (Cmax)
Description: The maximum measured concentration of hyoscine butylbromide in plasma.
Time Frame: Blood sampling within 2 hours prior to dosing, and 30, 60, and 120 minutes, and at 2.5, 3, 3.5, 3.75, 4, 4.25, 4.5, 5, 5.5, 6, 8, 12, 24, 36, 48 and 60 hours thereafter
Population: All subjects who had evaluable pharmacokinetic (PK) data for at least one of the treatment periods were included in the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram (pg)/millilitre (mL)
Groups:
- Buscopan® (REF): The subjects received the reference treatment (REF) which was 20 milligram (mg) of hyoscine butylbromide (trade name: Buscopan®, 2*10mg) which was administered as a single oral dose in the fasted state via a sugar coated tablet.
- Buscapina® (T): The subjects received the test treatment (T) which was 20 milligram (mg) of hyoscine butylbromide (trade name: Buscapina®, 2*10mg) which was administered as a single oral dose in the fasted state via a sugar coated tablet
Arm/Group | Buscopan® (REF) | Buscapina® (T)
Number analyzed (Participants) | 54 | 55
picogram (pg)/millilitre (mL) | 91 (93.4) | 80 (100.6)
Statistical Analysis 1: Comparison: Buscopan® (REF) vs Buscapina® (T); The study design is a two-stage Pocock-like group sequential design according to the alpha spending function approach. The alpha level for Stage 1 was 0.0377 (one-sided); Test type: Non-Inferiority or Equivalence — Bioequivalence of the test and reference product (for Stage 1) was assessed on the basis of the point estimate of the geometric mean ratio for Cmax in relation to the bioequivalence range of 80.00% to 125.00%; Geometric mean ratio (%): T/REF = 87.52, 92.46% CI 2-sided [77.18 to 99.24] — ANOVA model was used with 'sequence', 'treatment' and 'period' as fixed effects and 'subject within sequence' as a random effect after logarithmic transformation of the data

2. Primary Outcome: AUC Time Zero to Times of Last Quantifiable Concentration (AUC 0-t)
Description: Area under the concentration-time curve of hyoscine butylbromide in plasma over the time interval from 0 to the last quantifiable data point (AUC0-t).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)*pg/mL
Arm/Group | Buscopan® (REF) | Buscapina® (T)
Number analyzed (Participants) | 52 | 55
hour (h)*pg/mL | 807 (89.3) | 725 (89.1)
Statistical Analysis 1: Comparison: Buscopan® (REF) vs Buscapina® (T); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Bioequivalence of the test and reference products for Stage 1 was assessed on the basis of the 92.46% confidence intervals for the geometric mean (test/reference) ratio for the AUC0-t in relation to the bioequivalence range of 80.00% to 125.00%, with a one-sided alpha of 0.0377; Geometric mean ratio (%): T/REF = 91.74, 92.46% CI 2-sided [83.51 to 100.78] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve, With Extrapolation to Infinity (AUC0-∞).
Description: The area under the concentration-time curve of hyoscine butylbromide in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Buscopan® (REF) | Buscapina® (T)
Number analyzed (Participants) | 52 | 55
h*pg/mL | 847 (86.6) | 760 (88.5)
Statistical Analysis 1: Comparison: Buscopan® (REF) vs Buscapina® (T); The test product was compared to the reference product by means of statistical analysis; Test type: Superiority or Other; Geometric mean ratio (%): T/REF = 91.66, 92.46% CI 2-sided [83.59 to 100.51] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Area Under the Curve, for the Test Product, to the Time of the Maximum Concentration of the Reference Product and the Test Product (AUCReftmax)
Description: Area under the concentration-time curve of hyoscine butylbromide to the time of the maximum concentration of hyoscine butylbromide of the reference product (Buscopan®). This was calculated both for test and reference products.
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Buscopan® (REF) | Buscapina® (T)
Number analyzed (Participants) | 52 | 54
h*pg/mL | 187 (104.0) | 170 (121.8)
Statistical Analysis 1: Comparison: Buscopan® (REF) vs Buscapina® (T); The test product was compared to the reference product by means of statistical analysis; Test type: Superiority or Other; Geometric mean ratio (%): T/REF = 92.96, 92.46% CI 2-sided [81.94 to 105.47] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first administration of study medication to up to 96 hours of completion of the last period or up to 72 hours after withdrawal/withdrawing from the study (up to 34 days).
Arm/Group | Buscopan® (REF) | Buscapina® (T)
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

LIMITATIONS AND CAVEATS:
There was a stage 2 planned after stage 1 which was not performed as bioequivalence was concluded after completion of Stage 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property right.